CLINICAL TRIAL: NCT00809549
Title: Granulocyte-Colony Stimulating Factor In Ischemic Stroke (GIST): A Pilot Study
Brief Title: Study to Determine The Effect of a Drug Called Neupogen on Stroke Recovery
Acronym: GIST
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006076-01H
Record Dates: First submitted 2008-10-17; First posted 2008-12-17 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Ischemic Stroke
Keywords: Stroke; GCSF; Hematopoeitic; Neupogen; Filgrastim
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Filgrastim; pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Saline (Placebo Comparator)
  Interventions: Drug: Filgrastim
- Filgrastim (Experimental)
  Interventions: Drug: Filgrastim

INTERVENTIONS:
Drug: Filgrastim — 10 ug/kg sc once daily x 4 days. Repeated once, 6 weeks later.
  Other Names: Brand Name: Neupogen; rhG-CSF

SUMMARY:
1. Circulating bone marrow and blood vessel precursors home in to sites of ischemia and aid regeneration of injured tissue
2. Increasing the number of circulating precursors will improve in regeneration of damaged brain following ischemic stroke.

DETAILED DESCRIPTION:
We hypothesize that mobilization of bone marrow precursor cells into the blood stream will allow them to redistribute in the injured central nervous system and aid regeneration of damaged tissue. If the hypotheses is correct, it predicts that G-CSF treatment will improve the functional outcome of patients following acute ischemic stroke.

Underlying this work are the following considerations:

* Currently the clinical and functional outcomes following ischemic strokes are poor and require new treatment strategies.
* G-CSF administration is a well established routine treatment for the mobilization of hematopoietic and endothelial precursors from the bone marrow into the circulation.
* Acute ischemia locally increases factors that direct circulating bone marrow derived cells to home to these sites of injury.
* Evidence exists that bone marrow derived cells are able to repopulate different tissues including those of the CNS.
* Acute ischemic injury to the central nervous system provides a milieu for the regeneration of neural tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 45 and 85 years of age
* Patient is of either gender
* The qualifying stroke is ischemic with a total NIH Stroke Score less than 18.
* The stroke involves the non-dominant hemisphere including the cerebral cortex and results in hemiparesis. The inclusion of sub-cortical strokes will be permitted if the size is of 3 cm or greater. Patients suffering strokes involving the dominant hemisphere resulting in mild dysphasia are also eligible.
* The stroke is classified as a partial anterior cerebral syndrome by the Oxfordshire Criteria.
* NIHSS at baseline evaluation with:

  *Level of consciousness is not impaired as defined by an NIHSS between 0 and 1 on question 1a and
* Hemiparesis as defined by

  * an NIHSS between 1 and 4 on questions 5 and/or
  * an NIHSS between 1 and 4 on questions 6.
* Be able to start the experimental treatment a minimum of 3 days and a maximum of 10 days after the initial presentation with the stroke,
* Patient or surrogate gives informed consent,
* The patient is fluent in either French or English.

Exclusion Criteria:

* Patient with hemorrhagic stroke,
* Patients with a pre-morbid modified Rankin score > 2 (Appendix 3b),
* Patients with pre-morbid dementia by DSM-IV criteria.
* Patients with a known allergic reaction to G-CSF or a component of G-CSF.
* Patients with one or more significant co-morbidities expected to limit lifespan to less than 12 months. Examples include but are not limited to:

  * > CHF Class II NYHA
  * Known prior or ongoing malignancy except non-melanomatous skin cancer.
  * Acute or chronic infections (HIV, TB, etc.. )
  * Other significant cardiac, renal, hepatic or pulmonary dysfunction.
* Patients with organ dysfunction that would preclude tests required for this study. Examples include but are not limited to:

  *Serum Cr > 200 μmol/L that would prevent administration of contrast dye.
* Patients with a known history of bone marrow dysfunction, such as myeloid leukemia or myeloproliferative state that would prevent treatment with G-CSF.
* Patients with metal implants that would preclude MRI examination including but not limited to patients with

  * pacemakers,
  * ear implants, and
  * aneurysm brain clips.
* Patients with:

  * a history compatible with a thrombophilic state or
  * with a pre-existing known thrombophilic state.
* Patient unwilling or unable to comply with trial requirements.
* Patients with an ongoing history of illicit drug use.
* Female patients of child-bearing potential.
* Patients exposed to other investigational drugs in the last 3 months.
* Patients with known or suspected sickle cell disease,
* Patients with splenic enlargement or an illness that results in splenic enlargement (For example, but not limited to myeloproliferative syndromes, hairy cell leukaemia, malaria, hepatic cirrhosis…),
* Patients with an ongoing history of alcohol abuse,
* Patients with a known or suspected history of allergy to intravenous contrast agents used for CT scans,
* Patients that have received a chemotherapy agent within the previous 5 years (For example, but not limited to cyclophosphamide, anthracycline, methotrexate, fluorouracil…)
* Patients that have received a therapy within the previous 5 years that interferes with hematopoiesis or circulating blood cells (For example, but not limited to Lithium, Campath….)
* Patients that have received a cytokine within the last 6 months or are currently receiving a cytokine treatment (For example, but not limited to Erythropoietin, Granulocyte Macrophage Colony Stimulating Factor, Keratinocyte Growth Factor, Kit Ligand…)

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-07; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
A statistically significant increase in: mortality/ non-fatal grade III or greater adverse events measured by the NCI Common Toxicity Scale/ incidence of recurrent strokes/ worsening of neurological disabilities measured by standardized stroke scales. | 6 weeks, 3 months, 6 months and 12 months after the first dose of the study drug.

SECONDARY OUTCOMES:
The secondary endpoints address the feasibility and efficacy of the study treatment: adequacy of bone marrow cell mobilization/ validation of imaging sequences/ Identification of optimal parameters for follow-up to be used in a subsequent larger trial. | 6 weeks, 3 months, 6 months and 12 months after the first dose of the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sharma, MD, Principal Investigator — The Ottawa Hospital
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario